CLINICAL TRIAL: NCT05861960
Title: Endogenous Pain Modulation in Patients With Shoulder Arthroplasty for Osteoarthritis
Brief Title: Endogenous Pain Modulation Study
Acronym: EPM
Status: Recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-005-M
Record Dates: First submitted 2023-04-21; First posted 2023-05-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Osteo Arthritis Shoulders; Osteoarthritis Shoulder
Keywords: Total shoulder arthroplasty; Osteoarthritis; Quantitative sensory testing; Conditioned pain modulation; Temporal summation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Although most patients experience significant pain relief after total shoulder arthroplasty (TSA), pain persists for some patients even after surgery. The endogenous pain system may be involved in persisting postoperative pain in total knee arthroplasty (TKA) and total hip arthroplasty (THA) patients, but this has never been studies for TSA patients. Furthermore, psychological factors and coping strategies may also be of interest but have not yet been extensively studied in TSA patients.

Objective: The primary objective is to explore whether central sensitization and/or abnormal CPM responses are present in (a subgroup of) patients who will receive shoulder arthroplasty for osteoarthritis, and whether shoulder arthroplasty produces change in these measures of the endogenous pain modulatory system.

The secondary objective, in case patients with altered endogenous pain modulation are found, is to explore if change in pain over time, psychological factors and coping strategies differ between patients with and without altered pain modulation.

Study design: An exploratory prospective observational cohort study.

Study population: Patients (age 18 years or older) who are scheduled to undergo shoulder arthroplasty for osteoarthritis, at the Reinier Haga Orthopaedic Centre.

Intervention (if applicable): Not applicable.

Main study parameters/endpoints: The main study parameters are CPM and TS values at baseline and at 3 and 6 months after surgery, as well as the absence/presence of allodynia at baseline and at 3 and 6 months after surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden of participation will consist of completing questionnaires at baseline and at three and six months after surgery. In addition, subjects will undergo psychophysical testing at 3 moments, which can lead to redness or a burning sensation of the skin during the first 24 hours after testing. The investigators do not expect any additional risks associated with participation. There is no direct benefit for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs
* Scheduled to undergo primary total shoulder arthroplasty (TSA) or reversed shoulder arthroplasty (RSA) for primary shoulder osteoarthritis or cuff tear arthropathy
* American Society of Anesthesiologists score 1, 2 or 3
* Able to provide written informed consent

Exclusion Criteria:

* Regular use of anti-depressants or anti-epileptics for any purpose, including SNRIs and gabapentinoids
* The presence of any chronic pain disorder other than osteoarthritis
* Osteoarthritis in joints other than the affected shoulder, for which arthroplasty is/will be planned in the near future
* Difficulty with or inability to perform psychophysical testing (eg. in case of cognitive or psychiatric disorders)
* Difficulty with or inability to communicate with the investigators (eg. difficulty with the Dutch language, cognitive/memory disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are scheduled to undergo primary shoulder arthroplasty for shoulder osteoarthritis (OA) or rotator cuff tear arthropathy (CTA).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with adequate conditioned pain modulation (CPM, CPM value > 10%) | Before surgery
  The subjects will score pain perception during the stimuli using the electronic visual analogue scoring (eVAS) system. The eVAS is scored on a scale of 0 (no pain) to 10 (worst pain).
Percentage of patients with adequate conditioned pain modulation (CPM, CPM value > 10%) | 3 months
  The subjects will score pain perception during the stimuli using the electronic visual analogue scoring (eVAS) system. The eVAS is scored on a scale of 0 (no pain) to 10 (worst pain).
Percentage of patients with adequate conditioned pain modulation (CPM, CPM value > 10%) | 6 months
  The subjects will score pain perception during the stimuli using the electronic visual analogue scoring (eVAS) system. The eVAS is scored on a scale of 0 (no pain) to 10 (worst pain).
Percentage of patients with normal emporal summation (TS, TS value < 2 points) | Before surgery
  Subjects will verbally rate their pain during the test using the numeric rating scale (NRS). This is a scale on 0 (no pain) to 10 (worst pain).
Percentage of patients with normal emporal summation (TS, TS value < 2 points) | 3 months
  Subjects will verbally rate their pain during the test using the numeric rating scale (NRS). This is a scale on 0 (no pain) to 10 (worst pain).
Percentage of patients with normal emporal summation (TS, TS value < 2 points) | 6 months
  Subjects will verbally rate their pain during the test using the numeric rating scale (NRS). This is a scale on 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Mean pain score (NRS) | Before surgery, 3 months, 6 months
  Pain will be measured using the Numeric Rating Scal for pain (NRS). This is a scale on 0 (no pain) to 10 (worst pain).
Pain catastrophizing | Before surgery, 3 months, 6 months
  The Pain Catastrophizing Scale (PCS) is a 13-item questionnaire that assesses catastrophizing about pain. The total score ranges from 0-52. A score of 30 and higher indicates a clinically relevant level of catastrophizing.
Coping strategies | Before surgery, 3 months, 6 months
  The Brief COPE consists of 28 items, measuring 14 subscales. Each scale is measured by two items, with each item scoring form 1 to 4. Higher subscale scores indicate a higher use of that coping strategy.

OTHER OUTCOMES:
The number of complications | 3 months, 6 months
  The complications after surgery
Mean operating time | During surgery
  The operating time in mintues
Optimal/suboptimal positioning of the prothesis | Directly postoperatively
  The positioning of the prothesis categorized in optimal and suboptimal based on the regular x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Brechtje Hesseling, MSc, Principal Investigator — Reinier Haga Orthopedisch Centrum
Locations (1):
- Reinier Haga Orthopedic Center, Zoetermeer, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided